CLINICAL TRIAL: NCT06674902
Title: Short-term Effectiveness of High- and Low-intensity Percutaneous Electrolysis in Patients With Plantar Fasciitis
Brief Title: Electrolysis in Patients With Chronic Plantar Fasciitis
Acronym: Electrolysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Universidad Complutense de Madrid (Other); Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Sebastian Klich, Principle Investigator, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCM#2; #19/044 (Other: Clinical Ethics Committee of Hospital Clínico San Carlos)
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Plantar Fasciitis
Keywords: Pain; Electrolysis; shear-wave elastography; pain sensitivity
MeSH Terms: conditions — Fasciitis, Plantar; Pain

STUDY DESIGN:
Intervention Model Description: A triple-blinded, pilot randomized controlled trial
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 1: Electrolysis with 4 mA (Experimental): A charge of 24 mC will be delivered at 4 mA for 6 seconds, followed by a 54-second pause.
  Interventions: Device: Electrolysis Percutaneous Therapeutic (EPTE)
- Experimental 2: Electrolysis with 400 μA (Experimental): A charge of 24 mC will be delivered at 400 µA for 60 seconds.
  Interventions: Device: Electrolysis Percutaneous Therapeutic (EPTE)
- Experimental 3: Electrolysis with 600 μA (Experimental): A charge of 36 mC will be delivered at 600 µA for 60 seconds.
  Interventions: Device: Electrolysis Percutaneous Therapeutic (EPTE)

INTERVENTIONS:
Device: Electrolysis Percutaneous Therapeutic (EPTE) — EPTE device (Ionclinics, Valencia, Spain)

SUMMARY:
Aim of the Study

The aim of this study is to investigate the differential effects of high-intensity and low-intensity percutaneous electrolysis (PCE) on pain perception and muscle tissue properties in individuals with chronic plantar fasciitis.

Research Questions

Pain Perception:

Does high-intensity PCE induce greater changes in pressure pain threshold (PPT) in the plantar fascia compared to low-intensity PCE in individuals with chronic plantar fasciitis?

Muscle Tissue Properties:

Does high-intensity PCE reduce stiffness in the plantar fascia to a greater extent than low-intensity PCE in individuals with chronic plantar fasciitis?

DETAILED DESCRIPTION:
A randomized, controlled, triple-blind clinical trial will be conducted to compare the effects of a single session of percutaneous intertissued electrolysis in three different modes (two intervention groups with the same dose but different intensity and time parameters, and one intervention group with a different dose) in patients with chronic plantar fasciitis (PF).

This study will be conducted under the Consolidated Standards of Reporting Trials (CONSORT) guidelines for pragmatic clinical trials and the EQUATOR guidelines to improve health research quality and transparency. Since the study involves patients with plantar pain, participants' rights will be respected under the Declaration of Helsinki. The Ethics Committee of University Hospital 12 de Octubre must approve the study protocol before data collection begins. The study protocol will also be prospectively registered on ClinicalTrials.org before data collection begins.

Sociodemographic variables (age, sex, weight, height, and body mass index), clinical variables (pain intensity, disability related to PF, pain thresholds to pressure), mechanical variables (plantar fascia stiffness), and tolerance to the treatment (visual analog scale to assess the intensity of pain felt during the intervention) will be assessed. Sociodemographic variables will be collected before the intervention, clinical and mechanical variables before and after the intervention, and tolerance to treatment only after the intervention. The assessment of participants will be carried out by an assessor who will not know which intervention group the participant belongs to. Participants will not know what dose they received, and the physiotherapists performing the procedures will also not know what settings the electrotherapy device has.

Participants will be randomly assigned to one of three intervention groups using a random number generator (Research Randomizer, version 4.0). Individual cards with numbers assigned sequentially according to the randomization will be used, which will then be folded and placed in opaque, sealed envelopes to ensure the concealment of allocation. An external researcher will select the envelope and make the assignment, which will only be revealed to the external therapist setting the equipment parameters after the initial data collection is completed. The assessor, therapist, and participants will not know to which group they have been assigned.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older,
* unilateral heel pain lasting longer than 3 months,
* a clinical diagnosis of chronic plantar fasciitis according to the clinical practice guidelines of the Orthopaedic Section of the American Physical Therapy Association (APTA), i.e., sudden onset of pain on the plantar surface of the heel after a period of non-weight bearing, pain that is worse in the morning with the first step, and tenderness to palpation at the proximal attachment site of the plantar fascia.

Exclusion Criteria:

* previous lower extremity surgery,
* the presence of positive neurological signs consistent with nerve root compression,
* any medical conditions causing heel pain, such as rheumatoid arthritis, diabetes, or peripheral neuropathy,
* receipt of any foot treatment within the past 6 weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-11-11 (Estimated); Primary Completion 2024-11-22 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline, immediately after
  Participants will rate their pain intensity on an 11-point numeric rating scale (NPRS; 0 = no pain; 10 = worst possible pain). They will consider the pain intensity of their first step in the morning, the average pain intensity during the day, and the maximum pain experienced in the past week. The average of all these values will be used to calculate a pain intensity score for the primary analysis.

SECONDARY OUTCOMES:
Foot function | Baseline, immediately after
  Foot function will be assessed using the Foot Function Index (FFI), the most commonly used self-assessment tool for the foot. The FFI has been shown to be reliable, valid, and sensitive to change in individuals with chronic plantar heel pain.
  The Foot Function Index (FFI) consists of 23 self-reported questions divided into three subscales: pain (nine items), disability (nine items), and activity limitation (five items). Each item is rated on a 0-10 scale (0 = no pain or difficulty, 10 = worst possible pain or difficulty requiring help). Each subscale is scored as a percentage from 0% to 100%, with higher scores indicating lower function and poorer foot-related health-related quality of life. In this study, the total FFI score, calculated as the average of the three subscales, will be used for the primary analysis.
Pain threshold | Baseline, immediately after
  Participants will avoid pain meds/muscle relaxants for 24 hours. PPT will be measured using an electronic algometer at 30 kPa/s, with 3 measurements per site and a 30-second interval. PPT will be assessed bilaterally at the calcaneus, adjacent muscles, tibialis anterior, and a pain-free site. Inter-rater reliability: 0.74-0.97.
Tolerance | Baseline, during intervention, immediately after
  Participants will rate the intensity of pain experienced during the intervention on an 11-point numeric rating scale (NPRS; 0 = no pain; 10 = worst possible pain).
Tissue stiffness | Baseline, immediately after
  All images will be acquired using a General Electric Logiq P9 ultrasound system equipped with a linear 4-15 MHz probe, located in the Rehabilitation Department of the 12 de Octubre Hospital. Experienced researchers, with over 10 years of experience in musculoskeletal ultrasound and blinded to participant group assignment, will perform the imaging. Device parameters will be identical for all measurements (gain 55 dB, dynamic range 85, brightness 17, depth 4 cm, frequency 8 MHz). The plantar fascia image will be acquired in a longitudinal plane. Subsequently, shear wave elastography mode will be activated, and a region of interest 1 cm wide (corresponding to the width of the algometer head) and an appropriate height to analyze the entire thickness of the fascia will be marked. The ultrasound system will automatically calculate tissue stiffness parameters within the marked region (shear wave velocity and Young's modulus).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Valera-Calero, Study Director — Universidad Complutense de Madrid
Locations (1):
- Faculty of Nursery, Physiotherapy and Podiatry, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alburquerque-Sendin F, Rios-Leon M, Valera-Calero JA, Plaza-Manzano G, Fernandez-de-Las-Penas C, Ortega-Santiago R, Priscila Rodrigues-de-Souza D. Clinical, Psychological, and Neurophysiological Outcomes Associated with Pain and Function in Individuals with Unilateral Plantar Heel Pain. Pain Med. 2022 Aug 31;23(9):1613-1620. doi: 10.1093/pm/pnac018. PMID 35089360
- [Background] Rios-Leon M, Valera-Calero JA, Ortega-Santiago R, Varol U, Fernandez-de-Las-Penas C, Plaza-Manzano G. Analyzing the Interaction between Clinical, Neurophysiological and Psychological Outcomes Underlying Chronic Plantar Heel Pain: A Network Analysis Study. Int J Environ Res Public Health. 2022 Aug 18;19(16):10301. doi: 10.3390/ijerph191610301. PMID 36011936
- [Background] Valera-Calero JA, Sanchez-Mayoral-Martin A, Varol U. Short-term effectiveness of high- and low-intensity percutaneous electrolysis in patients with patellofemoral pain syndrome: A pilot study. World J Orthop. 2021 Oct 18;12(10):781-790. doi: 10.5312/wjo.v12.i10.781. eCollection 2021 Oct 18. PMID 34754834